CLINICAL TRIAL: NCT05671419
Title: Mindful Self-Compassion for Anxiety Disorders and Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Elizabeth Hoge, Professor of Psychiatry, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0005683
Record Dates: First submitted 2022-12-31; First posted 2023-01-04 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Anxiety Disorders; Generalized Anxiety Disorder; Social Anxiety Disorder; Social Phobia; Panic Disorder; Agoraphobia; Major Depressive Disorder
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder; Phobia, Social; Panic Disorder; Agoraphobia; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The study investigator will be masked to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Self-Compassion (Experimental): Mindful Self-Compassion (MSC) is a weekly class given for 8 weeks. The individual classes last about 2 hours each. The class is provided in a group setting.
  Interventions: Behavioral: Mindful Self-Compassion
- Treatment as Usual (TAU) (No Intervention): The TAU arm will not receive the additional treatment from the study. Subjects will receive psychiatric treatment from their usual providers.

INTERVENTIONS:
Behavioral: Mindful Self-Compassion — The course teaching mindfulness meditation skills relevant to cultivating self-compassion.
  Arms: Mindful Self-Compassion

SUMMARY:
The study will compare 8-week Mindful Self-Compassion training, compared to a control group that does not receive the intervention, on anxiety and depression symptom severity in patients with diagnosed anxiety disorders (generalized anxiety disorder, social anxiety disorder, and panic disorder) or major depressive disorder.

DETAILED DESCRIPTION:
Anxiety disorders, such as generalized anxiety disorder, social anxiety disorder, and panic disorder, and depressive disorders result in significant distress, impairment in social and occupational functioning and increased risk for suicide. While there are medication and psychotherapy treatment options, they can sometimes be difficult to access and may be ineffective for a proportion of the population. Also, many patients are reluctant to take psychiatric medication, and many prefer to avoid psychiatric care altogether due to stigma or distrust of medical care settings such as a psychiatry clinic. Mindfulness meditation training can be provided outside of a medical care setting and may be more acceptable and feasible for some patients.

One way that mindfulness meditation may provide unique benefits for anxiety and depression is through decreasing self-judgment and increasing self-compassion. Research has shown that people with anxiety disorders, for example, have lower levels of self-compassion than people without anxiety. This is consistent with theories about the development and phenomenology of anxiety disorders, which are characterized as having high levels of self-criticism. Mindfulness-based interventions have been shown to improve self-compassion and self-acceptance.

In this study, patients with anxiety disorders or depression will be randomized to either an 8-week class called Mindful Self-Compassion training or a group that does not receive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have a primary anxiety disorder (social anxiety disorder, generalized anxiety disorder, panic disorder, or agoraphobia) or major depressive disorder, current
* Must score low on self-compassion, as measured by the self-compassion scale
* Must understand study procedure and willing to participate in all testing visits, and treatment as assigned
* must be able to give informed consent to the study procedures

Exclusion Criteria:

* Comorbid psychiatric disorder other than anxiety or depression, such as psychotic disorder, obsessive compulsive disorder, eating disorders (i.e., anorexia and bulimia), bipolar disorder; developmental or organic mental disorders; and current (past 6 months) substance use disorders and current post-traumatic stress disorder as assessed by clinician at screening visit
* A serious medical condition that may result in surgery or hospitalization.
* A history of head trauma causing prolonged loss of consciousness, or ongoing cognitive impairment
* Inability to understand study procedures or informed consent process, or significant personality dysfunction likely to interfere with study participation (assessed during the clinical interview).
* Subjects who will be non-compliant with the study procedures. This may include planned travel out of town.
* Subjects taking some psychiatric medication such as barbiturates or antipsychotics. Sleep medications and some anti-depressants will be allowed, if the subject has been taken at stable dose 8 weeks prior to baseline and the patient plans to continue at the same dose through the trial.
* Concurrent psychotherapy initiated within 1 month of screen interview, or ongoing psychotherapy of any duration directed specifically toward the treatment of anxiety (such as Cognitive Behavioral Therapy).
* Individuals who have completed a course of MSC or an equivalent meditation training in the last year.
* Individuals reporting significant active suicidal ideation or suicidal behaviors within the past year.
* Individuals with a medical condition (i.e., epilepsy) that may be exacerbated by study treatment, as determined by a study physician or nurse practitioner based on history, physical, and/or labs.
* Adults unable to consent
* Pregnant women
* Prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | 8 weeks
  Self-report questionnaire of anxiety and depression symptoms, 14 items using 4-point likert scale

SECONDARY OUTCOMES:
Self-compassion Scale | 8 weeks
  Self-Report questionnaire of 26 items on 5 point likert scale
Liebowitz Social Anxiety Scale - Self-Report | 8 weeks
  Measures severity of social anxiety
PROMIS-Anxiety-Short form | 8 weeks
  measures anxiety symptoms using HealthMeasures system
PROMIS-Depression-Short Form | 8 weeks
  measures depression symptoms using HealthMeasures system

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hoge, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Individual-level participant data collected will not be made available to the general public due to conditions of ethical approval regarding confidentiality.